CLINICAL TRIAL: NCT01356628
Title: A Phase II Study of PD-0332991 in Adult Patients With Advanced Hepatocellular Carcinoma
Brief Title: A Clinical Research Study to Determine Whether PD 0332991 May Be Effective in Treating Patients With Liver Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Cancer Center at Thomas Jefferson University (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Organization: Thomas Jefferson University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11D.14; JT 1848 (Other: JeffTrial Number)
Record Dates: First submitted 2011-05-10; First posted 2011-05-19 (Estimated); Results first posted 2018-01-05 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Advanced Hepatocellular Carcinoma; HCC; Liver Cancer
Keywords: Advanced Hepatocellular Carcinoma; HCC; Liver Cancer; PD-0332991
MeSH Terms: conditions — Liver Neoplasms | interventions — palbociclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- PD-0332991 (Experimental): PD-0332991 in the Treatment in Patients with Advanced Hepatocellular Carcinoma
  Interventions: Drug: PD-0332991

INTERVENTIONS:
Drug: PD-0332991 — PD-0332991, 125mg, 3 cycles

SUMMARY:
This is a Phase 2 Study of PD-0332991 in the treatment of patients with Advanced Hepatocellular Carcinoma (HCC), a type of adenocarcinoma and the most common type of liver tumor. PD-0332991 is a compound that stops the tumor cell from entering the Synthesis phase of the cell cycle, therefore stopping DNA multiplication and decreased tumor cell copying.

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) is the fifth most common cancer worldwide and the third most frequent cause of cancer-related mortality. To date, surgical resection and liver transplantation are considered the main curative treatment options for HCC (El-Serag et al. 2006). However, the majority (~75%) of patients present with advanced tumor stage and poor liver function, rendering the patient ineligible for surgical interventions. Until the multikinase inhibitor sorafenib (Nexavar) was approved for the treatment of HCC in patients with unresectable disease (disease that can't be removed by surgery), there were no standard systemic therapies, as classical cell killing drugs (administered singularly or in combination) had not led to reproducible response rates or survival benefit. Despite this, response rates to sorafenib are low with overall benefits modest, and moreover the toxicity profile of the drug limits treatment for many patients. There is still a critical need for additional effective drugs to treat advanced HCC.

PD-0332991 is an orally available, selective inhibitor of cyclin-dependent kinase 4/6 (CDK4/6), a key regulator of cell growth. Pre-clinical data with PD-0332991 demonstrated potent target-specificity. PD-0332991 demonstrated significant inhibition of tumor cell growth in hepatoma cell lines, as well as animal and xenograft model systems, and was more effective than the currently approved drug, sorafenib in these systems. Initial clinical trials have demonstrated and acceptable toxicity profile for the drug. Thus, PD-0332991 represents an ideal candidate for the treatment of patients with advanced HCC.

This trial is an open-label non-randomized single-institution study for subjects with inoperable, recurrent/refractory, advanced hepatocellular carcinoma (HCC). Subjects must have failed or be intolerant of standard first line therapy, sorafenib (Nexavar®). Eligible subjects will receive 125 mg PD-0332991 capsules orally once daily, administered on days 1-21 of a 28-day cycle, in repeated cycles. The primary objective of the study is to assess the time to disease progression (TTP). Secondary objectives include assessment of safety and tolerability, and determination of overall survival (OS) and response rate (RR).

Subjects will be permitted to receive protocol directed therapy until disease progression as determined by modified RECIST (Response Evaluation Criteria in Solid Tumors) guidelines or clinical progression, unacceptable toxicity, withdrawal of consent or death. Tumor response assessment will be performed by the Investigator and will consist of evaluation by CT or MRI every 8 weeks. Subjects who discontinue therapy will still be followed for safety on Day 28 (± 3 days), Day 56 (± 3 days) and every 3 months thereafter from the last administration of protocol-directed therapy or until death.

Subjects will be continuously assessed for evidence of acute and cumulative toxicity. Vital signs, physical examinations, performance status, laboratory safety tests will be obtained and assessed prior to drug administration at regular intervals throughout the study. Toxicity will be evaluated every 2 weeks during the first 3 cycles and thereafter monthly (once per cycle) by the Investigator according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), Version 4.0.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, age > or = 18 years with HCC refractory to currently available therapies.
2. Documented HCC by at least 2 out of 3 mentioned criteria and evidence of non-resectability by a multidisciplinary team:

   A. Radiological - MRI with arterial enhancement and rapid venous washout B. Biopsy C. Serum alpha-fetoprotein level > or = 200
3. Positive staining for RB-function on tumor biopsy.
4. Subject must be able to give written informed consent and be able to follow protocol requirements
5. Life expectancy greater than 3 months
6. Be Child's-Pugh class A or B
7. ECOG Performance status of < or = 2
8. If female of childbearing potential must have negative pregnancy test at screening and may not be breast-feeding
9. Females of child-bearing potential (< one year post-menopausal with documented FSH greater than 30 IU/L or surgically not sterile), must agree to practice an effective method of avoiding pregnancy (including oral or implanted contraceptives, intrauterine device, condom, diaphragm with spermicidal, cervical cap, abstinence or sterile sex partner) from the time informed consent is signed through follow-up. Males must agree to take appropriate precautions to avoid fathering a child from screening through follow-up.
10. No other active malignancy requiring treatment in the last 3 years other than adequately treated non-melanomatous skin cancer, adequately treated cervical carcinoma in-situ, superficial adequately treated bladder cancer or prostatic intraepithelial neoplasia without evidence of prostate cancer.
11. Adequate bone marrow, liver and renal function as assessed by the following:

    A. Hemoglobin > or = 8 g/dL B. WBC > or = 4,000/uL C. Absolute neutrophil count > or = 1,500/uL D. Platelets > or = 75,000/uL E. Total bilirubin < or = 1.5 times ULN F. ALT and AST < or = 5 times ULN G. Creatinine < or = 1.5 times ULN H. Albumin > or = 2.5 mg/dL
12. Subjects who have received previous radiotherapy, loco-regional, or systemic therapy are eligible. A minimum interval of 4 weeks since the last anti-cancer treatment of any kind is required.
13. Subjects with brain metastases or a history of previously treated brain metastasis are eligible but must:

A. Have been treated by surgery or stereotactic radiosurgery (SRS) at least 4 weeks prior to enrollment B. AND have a baseline MRI or CT that shows no evidence of active intercranial disease C. AND be off steroids for at least 1 week prior to study enrollment

Exclusion Criteria:

1. Any concurrent active malignancy requiring treatment (other than basal or squamous cell carcinoma of the skin, carcinoma in situ of the cervix, superficial bladder tumors, or other malignancies curatively treated > 3 years prior to study entry)
2. History of severe cardiovascular disease within the last 12 months: symptomatic congestive heart failure, myocardial infarction, coronary artery disease (CAD), life threatening arrhythmias, uncontrolled hypertension
3. Renal failure requiring hemo- or peritoneal dialysis
4. Unstable systemic diseases or active uncontrolled infection
5. Known history of HIV infection
6. Clinically significant gastrointestinal bleeding within 30 days prior to study entry
7. Major surgery, open biopsy or significant traumatic injury within 4 weeks prior to study entry
8. Child's-Pugh Class C
9. Any malabsorption problem that, in the investigator's opinion, would prevent adequate absorption of the study drug
10. Presence of any other medical complications that in the investigator's opinion, suggests a survival of < 3 months
11. Substance abuse, or medical, psychological or social conditions that may interfere with the patient's participation in the study or evaluation of the study results
12. Patient inability to swallow oral medications
13. Any condition that is unstable or which could jeopardize the safety of the patient and his/her compliance in the study
14. Pregnant or breast-feeding patients
15. Being of reproductive potential and unable or unwilling to practice an effective contraceptive method
16. Lack of positive staining for RB-function on tumor biopsy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2011-05-25 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-12-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Avnish Bhatia, MD, Principal Investigator — Sidney Kimmel Cancer Center at Thomas Jefferson University
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Fry DW, Harvey PJ, Keller PR, Elliott WL, Meade M, Trachet E, Albassam M, Zheng X, Leopold WR, Pryer NK, Toogood PL. Specific inhibition of cyclin-dependent kinase 4/6 by PD 0332991 and associated antitumor activity in human tumor xenografts. Mol Cancer Ther. 2004 Nov;3(11):1427-38. PMID 15542782
- [Background] Toogood PL, Harvey PJ, Repine JT, Sheehan DJ, VanderWel SN, Zhou H, Keller PR, McNamara DJ, Sherry D, Zhu T, Brodfuehrer J, Choi C, Barvian MR, Fry DW. Discovery of a potent and selective inhibitor of cyclin-dependent kinase 4/6. J Med Chem. 2005 Apr 7;48(7):2388-406. doi: 10.1021/jm049354h. PMID 15801831
- [Background] Rivadeneira DB, Mayhew CN, Thangavel C, Sotillo E, Reed CA, Grana X, Knudsen ES. Proliferative suppression by CDK4/6 inhibition: complex function of the retinoblastoma pathway in liver tissue and hepatoma cells. Gastroenterology. 2010 May;138(5):1920-30. doi: 10.1053/j.gastro.2010.01.007. Epub 2010 Jan 25. PMID 20100483
- See also: Thomas Jefferson University Hospitals — http://www.JeffersonHospital.org/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | PD-0332991
Started | 23
Completed | 23
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | PD-0332991
Number analyzed (Participants) | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 22
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 7
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 12
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 23

OUTCOME MEASURES:

1. Primary Outcome: Time to Disease Progression
Description: Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST Version 1.1), as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). The appearance of one or more new lesions is also considered progression.
Time Frame: From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
Measure: Mean (Full Range); unit: months
Arm/Group | PD-0332991
Number analyzed (Participants) | 23
months | 8 [3 to 8]

2. Secondary Outcome: Number of Adverse Events
Description: The number and nature of adverse events as a measure of safety and tolerability. Safety analysis will be conducted on all patients who receive at least one dose of PD-0332991 during the study period or follow-up. An adverse event is any unfavorable and unintended sign, symptom, syndrome or illness that develops during the period of observation in the clinical study, including a new illness or condition, worsening of a concomitant illnesses or condition, effect of the study medication or combination of 2 or more factors.
Time Frame: From date of randomization through study completion, assessed up to 100 months
Measure: Number; unit: Adverse Events
Arm/Group | PD-0332991
Number analyzed (Participants) | 23
Adverse Events | 504

3. Secondary Outcome: Overall Survival (OS)
Description: Overall survival (OS) is measured from the entry onto the trial until death of any cause. Date and cause of death will be recorded. The cause of death will be categorized as either cancer-related or cancer-unrelated.
Time Frame: Every 2 weeks during first 3 cycles, then monthly during treatment. Then Day 28, Day 56 and every 3 months from last administration of protocol directed therapy or death
Population: excluding 2 patients who are alive at 137 and 73 weeks.
Measure: Median (Full Range); unit: weeks
Arm/Group | PD-0332991
Number analyzed (Participants) | 23
weeks | 40 [24 to 96]

4. Secondary Outcome: Response Rate (RR)
Description: The best overall response is the best response recorded from the start of treatment until disease progression or recurrence. The objective response rate is the proportion of subjects with either a confirmed complete response (CR) or a confirmed partial response (PR) as determined using modified RECIST (Response Evaluation Criteria In Solid Tumors) criteria. Subjects with the response of stable disease (SD) will be recorded and documented. Disease control rate defined as CR+PR+SD will be calculated for all subjects treated with PD-0332991.
Time Frame: Every 8 weeks
Population: 4 patients were non-evaluable
Measure: Count of Participants; unit: Participants
Arm/Group | PD-0332991
Number analyzed (Participants) | 19
Participants
  Partial Response (PR) | 1
  Complete Response (CR) | 0
  Stable Disease (SD) | 7
  Progressive Disease | 11

ADVERSE EVENTS:
Time Frame: The adverse event reporting period for this trial begins when the patient receives the first dose of investigational medication and ends 28 days after the patient receives the last dose of his/her study medication regimen for all non-serious adverse events. All serious adverse events will be followed through safety follow-up visits until resolution or return to baseline condition.
Description: adverse medication reactions such as overdose, abuse, withdrawal, sensitivity, or toxicity; unrelated illnesses, worsening of a preexisting illness; Injury, accidents, abnormalities in physiological testing or physical examinations, Laboratory abnormalities
Arm/Group | PD-0332991
All-Cause Mortality (participants affected / at risk) | 20/23
Serious Adverse Events (participants affected / at risk) | 11/23
Other Adverse Events (participants affected / at risk) | 23/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PD-0332991 (N=23)
Vomiting (Gastrointestinal disorders) | 2 (2)
Peritoneal Infection (Gastrointestinal disorders) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 3 (3)
Neutropenia (Blood and lymphatic system disorders) | 3 (4)
Lower abdomen pain (Gastrointestinal disorders) | 3 (3)
Lower leg weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Spinal cord compression (Nervous system disorders) | 1 (1)
Hyperbilirubinema (Blood and lymphatic system disorders) | 3 (4)
Fever (Infections and infestations) | 1 (1)
Hypercalcemia (Blood and lymphatic system disorders) | 1 (1)
Hyperkalemia (Blood and lymphatic system disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2)
Fracture of left Humorous (General disorders) | 1 (1)
Dehydration (General disorders) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1)
Lower Gastrointestinal Hemorrhage (Gastrointestinal disorders) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Hepatic Failure (Hepatobiliary disorders) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PD-0332991 (N=23)
Thrombocytopenia (Blood and lymphatic system disorders) | 20 (56)
Alanine Aminotransferase Increased (Blood and lymphatic system disorders) | 10 (28)
Alkaline Phosphate Increase (Blood and lymphatic system disorders) | 8 (15)
Anemia (Blood and lymphatic system disorders) | 13 (23)
Anorexia (Psychiatric disorders) | 7 (9)
Ascites (Renal and urinary disorders) | 10 (22)
Aspartate Aminotransferase Increased (Blood and lymphatic system disorders) | 5 (8)
Blood in Stool (Gastrointestinal disorders) | 2 (2)
Blurred Vision (Eye disorders) | 3 (3)
Body Aches/Pan (General disorders) | 7 (8)
Chills (General disorders) | 3 (5)
Cirrhosis (Renal and urinary disorders) | 3 (4)
Cold (General disorders) | 6 (9)
Constipation (Gastrointestinal disorders) | 1 (2)
COPD (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Creatine increase (Blood and lymphatic system disorders) | 5 (7)
Decreased Appetite (Metabolism and nutrition disorders) | 2 (5)
Delirium, Post-Op (Psychiatric disorders) | 2 (4)
Depression (Psychiatric disorders) | 4 (14)
Diabetes (Blood and lymphatic system disorders) | 5 (9)
Diarrhea (Gastrointestinal disorders) | 5 (10)
Diverticulitis (Gastrointestinal disorders) | 4 (9)
Dizzyness (General disorders) | 4 (7)
Dry cracked palms (Skin and subcutaneous tissue disorders) | 3 (6)
Dysphasia (Nervous system disorders) | 1 (1)
Dyspnea (Reproductive system and breast disorders) | 1 (1)
Edema (General disorders) | 10 (13)
Emesis (Gastrointestinal disorders) | 4 (6)
Epigastric (Gastrointestinal disorders) | 3 (4)
Epistaxis (General disorders) | 2 (3)
Fall (General disorders) | 6 (6)
Fatigue (General disorders) | 1 (1)
Fever (Infections and infestations) | 2 (3)
Fungal Esophageal Infection (Infections and infestations) | 3 (5)
Gas (Gastrointestinal disorders) | 1 (1)
Gas reflex (General disorders) | 3 (3)
GERD (Gastrointestinal disorders) | 2 (2)
GI Bleeding (Gastrointestinal disorders) | 6 (7)
Gout (General disorders) | 1 (1)
Heartburn (Gastrointestinal disorders) | 3 (4)
Hepatitis C (Infections and infestations) | 1 (3)
Hyperbilirubinema (Blood and lymphatic system disorders) | 3 (5)
Hypercalemia (Blood and lymphatic system disorders) | 3 (4)
Hyperglycemia (Blood and lymphatic system disorders) | 5 (8)
Hyperkalemia (Blood and lymphatic system disorders) | 2 (3)
Hyperlipidemia (Blood and lymphatic system disorders) | 4 (5)
Hypermagnesemia (Blood and lymphatic system disorders) | 1 (1)
Hypertension (Blood and lymphatic system disorders) | 2 (3)
Hypoalbuminemia (Blood and lymphatic system disorders) | 4 (5)
Hyponatremia (Blood and lymphatic system disorders) | 3 (4)
Hypocalcemia (Blood and lymphatic system disorders) | 4 (6)
Hypokalemia (Blood and lymphatic system disorders) | 1 (1)
Hypomagnesemia (Blood and lymphatic system disorders) | 4 (10)
Hypophosphatemia (Blood and lymphatic system disorders) | 2 (2)
Hypotension (Blood and lymphatic system disorders) | 3 (4)
Increase in Creatine (Blood and lymphatic system disorders) | 3 (3)
Infection, C.Diff (Infections and infestations) | 2 (2)
Inguinal hernia (Gastrointestinal disorders) | 3 (8)
Injection Site Reaction (General disorders) | 1 (1)
INR increased (Blood and lymphatic system disorders) | 1 (1)
Insomnia (Nervous system disorders) | 5 (9)
Jaundice (Renal and urinary disorders) | 1 (1)
leg pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 5 (9)
Lightheadedness (General disorders) | 1 (1)
Low ANC (Blood and lymphatic system disorders) | 3 (7)
Lymphocytopenia (Blood and lymphatic system disorders) | 2 (5)
Mucositis (Gastrointestinal disorders) | 4 (4)
Muscle cramping (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (2)
Nausea (General disorders) | 5 (14)
Neck Fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Neuropathy (Nervous system disorders) | 6 (8)
Neutropenia (Blood and lymphatic system disorders) | 2 (2)
Night Sweats (General disorders) | 2 (2)
Pain (General disorders) | 3 (4)
Polymicrobial Bacteremia (Infections and infestations) | 1 (1)
Pruritus (Itching) (Skin and subcutaneous tissue disorders) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 2 (2)
Rash Pustular (Skin and subcutaneous tissue disorders) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1)
Sleep Apnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Stomach Virus (Gastrointestinal disorders) | 1 (1)
Taste Alteration (Nervous system disorders) | 1 (1)
Tonsillectomy (Surgical and medical procedures) | 1 (2)
Urinary Frequency and burning (Renal and urinary disorders) | 1 (1)
Urine Discoloration (Renal and urinary disorders) | 1 (1)
Vision Change (Eye disorders) | 1 (2)
Weakness (General disorders) | 1 (1)
ANC decreased (Blood and lymphatic system disorders) | 1 (2)
Dry Skin (Skin and subcutaneous tissue disorders) | 1 (1)
Metabolism and nutrition disorder (Metabolism and nutrition disorders) | 1 (1)
Neoplasm benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cramping hands and legs (Musculoskeletal and connective tissue disorders) | 1 (2)
Hemorrhoids (Gastrointestinal disorders) | 1 (1)
Emphesyma (Respiratory, thoracic and mediastinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-01): https://cdn.clinicaltrials.gov/large-docs/28/NCT01356628/Prot_SAP_000.pdf